CLINICAL TRIAL: NCT00132860
Title: Antibiotic Treatment of Patients With Chronic Obstructive Lung Disease: A Prospective, Randomized, Double-Blind Placebo-Controlled Study of Intermittent, Prophylactic Antibiotic Treatment With Azithromycin
Brief Title: Prophylactic Antibiotic Treatment of Patients With Chronic Obstructive Lung Disease (COLD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ProToCOL
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2005-10-19 (Estimated); Status verified 2005-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

INTERVENTIONS:
Drug: azithromycin

SUMMARY:
The purpose of the study is to investigate, in patients with moderate to severe chronic obstructive lung disease, whether intermittent antibiotic treatment leads to:

* A slower rate of decline in forced expiratory volume in one second (FEV1);
* A reduction in the frequency and severity of exacerbations;
* Fewer hospital admissions for chronic obstructive pulmonary disease (COPD);
* Lower mortality;
* An improved quality of life as compared to a group of placebo treated patients.

DETAILED DESCRIPTION:
Study Population: Patients with moderate to severe chronic obstructive lung disease.

Trial Phase: IV

Study Design: Prospective, randomised, double-blind, placebo- controlled clinical trial.

Study Medicine: Azithromycin.

Drug Administration: Oral.

Drug Dose: 500 mg once daily for 3 days every month.

Duration of Treatment: 3 years

Number of Evaluable Patients: 200 per treatment arm

Number of Included Patients: 400 per treatment arm, 800 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 50 years of age, with a current admission for exacerbation of COLD or at least one admission within the previous two years.
* Current or ex-smoker
* Postbronchodilator FEV1 < 60% in stable condition (> 4 weeks after hospitalisation)
* < 300 ml bronchodilator reversibility in FEV1

Exclusion Criteria:

* Patients with end-stage COLD, who are not expected to survive for 3 years (typically bedridden patients being dyspnoeic in rest).
* Patients with known other respiratory tract infection, e.g. tuberculosis or aspergillosis, in whom the intervention is known to be inefficient.
* Patients with pulmonary malignancy
* Patients with other pulmonary diseases than COLD.
* Patients with immunodeficiency. However, COLD patients treated with steroids can be included.
* Patients with known hereditary disposition to lung infections such as alfa-1-antitrypsin deficiency, cystic fibrosis or primary ciliary dyskinesia.
* Patients receiving longterm antibiotic treatment ( e.g. recurrent cystitis).
* Patients with known allergy or intolerance to azithromycin
* Pregnant or breastfeeding women
* Manifest heart, liver or renal insufficiency
* Patients that, for reasons not stated above, are unlikely to be able to participate in a study period of 3 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2001-05; Study Completion 2007-12

PRIMARY OUTCOMES:
change in postbronchodilator FEV1

SECONDARY OUTCOMES:
number of hospital admissions and number of hospital days
mortality
quality of life
use of medication
prevalence of respiratory pathogens
prevalence of macrolide resistance
inflammatory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Svend S Pedersen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Sorensen AK, Holmgaard DB, Mygind LH, Johansen J, Pedersen C. Neutrophil-to-lymphocyte ratio, calprotectin and YKL-40 in patients with chronic obstructive pulmonary disease: correlations and 5-year mortality - a cohort study. J Inflamm (Lond). 2015 Mar 18;12:20. doi: 10.1186/s12950-015-0064-5. eCollection 2015. PMID 25908927
- [Derived] Holmgaard DB, Mygind LH, Titlestad IL, Madsen H, Pedersen SS, Johansen JS, Pedersen C. Plasma YKL-40 and all-cause mortality in patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2013 Dec 30;13:77. doi: 10.1186/1471-2466-13-77. PMID 24373580